CLINICAL TRIAL: NCT04326231
Title: Cognoa ASD Digital Therapeutic Engagement and Usability Study
Brief Title: Cognoa Autism Spectrum Disorder (ASD) Digital Therapeutic Engagement and Usability Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID and the Study was withdrawn (limited recruitment within study timeline)
Sponsor: Cognoa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PRO-003
Record Dates: First submitted 2020-03-23; First posted 2020-03-30 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cognoa ASD Therapeutic Device (Experimental): Usability assessment of Cognoa ASD Therapeutic Device
  Interventions: Device: Usability assessment of Cognoa ASD Therapeutic Device

INTERVENTIONS:
Device: Usability assessment of Cognoa ASD Therapeutic Device — Usability assessment of Cognoa ASD Therapeutic Device

SUMMARY:
Cognoa will measure usability, engagement with the device, and changes in parent-reported socialization during a 4-week period of intervention at home with the Cognoa ASD therapeutic device.

DETAILED DESCRIPTION:
Parents who consent will be given access to the study device through its caregiver and child-facing smartphone app that provides therapeutic content. In order to access the study device app, parents will be provided access to two other apps. The first is Testflight. TestFlight is an online service for over-the-air installation and testing of mobile applications, currently owned by Apple Inc.that allows users to test iOS apps before they are released to the App Store. Parents will also be provided access to the Cognoa for Child Development app in order to create an account as a means to gain access to the study device app. The parents will only be able to engage with the study device app once they have created an account in the Cognoa for Child for Development app

ELIGIBILITY:
Inclusion Criteria:

* Functional English language capability in the home environment.
* Parent, Guardian, or legal authorized representative (LAR) must be able to read, understand and sign the Informed Consent Form (ICF)
* Female or Male, > 3 to < 9 years of age and parent/caregiver
* Diagnosis of Autism Spectrum Disorder, within the last 12 months
* Parent, Guardian, or legal authorized representative (LAR) must have smartphone capabilities for downloading Testflight software; test versions of the Cognoa for Child development app; and test versions of the Cognoa Digital Therapeutic app (iOS 12.0 and up and Apple iPhone 8 and higher)

Exclusion Criteria:

* Participants with any other medical, behavioral, or developmental condition that in the opinion of the investigator may confound study data/assessments.
* Participants with planned extensive travel (more than 1 week) during the course of the 4 week intervention time period.
* Participants with deafness or blindness.
* Participants with known physical impairments affecting their ability to use their hands.
* Participants with active diagnosis of epilepsy and uncontrolled seizures.
* Participants whose age on the date of enrollment is outside the target age range

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Abrams, PhD, Principal Investigator — Cognoa, Inc.
Locations (1):
- Cognoa, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Withdrawn (limited recruitment within study timeline)
Pre-assignment Details: The protocol enrollment number represents Child/Caregiver enrollment in the study.
Period: Overall Study
Arm/Group | Cognoa ASD Therapeutic Device
Started (10 subjects represents Child/Caregiver pair) | 10 (Child/Caregiver pair)
Completed (10 subjects represents Child/Caregiver pair) | 0 (COVID Withdrawn)
Not Completed | 10
Not completed — COVID Withdrawn (limited recruitment within study timeline) | 10

BASELINE CHARACTERISTICS:
Population: Up to 30 caregivers and children diagnosed with ASD ages > 3 to < 9 years of age will be recruited from across the U.S.
  Baseline data was only collected for children. This study was terminated data was not collected.
  Zero participants completed the study due to COVID.
Groups:
- Cognoa ASD Therapeutic Device: Usability assessment of Cognoa ASD Therapeutic Device Usability assessment of Cognoa ASD Therapeutic Device: Usability assessment of Cognoa ASD Therapeutic Device
Arm/Group | Cognoa ASD Therapeutic Device
Number analyzed (Participants) | 0
Age, Categorical — Study was terminated and data was not collected.
Sex: Female, Male — Study was terminated and data was not collected.
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants] — Study was terminated and data was not collected.

OUTCOME MEASURES:

1. Primary Outcome: Vineland Adaptive Behavior Scales, Third Edition
Description: Change was calculated on an average from all relevant time points used in the calculation in the Time Frame ( baseline assessment, 4 weeks of intervention 4-6 times a week, weekly surveys of usability, final assessment); These measures were not completed due to COVID
  Change in scores on the Vineland-3 domain level caregiver report social skills and relationships, measures of usability.
  Qualitative descriptors: scores of 1 to 17 may be considered Average, 18 to 20 Elevated, and 21 to 24 Clinically Significant
  Caregivers partially completed their scores on the Vineland Adaptive Behavior Scales, Third Edition, This was due to COVID and not being able to complete the study.
  0 Caregivers had their scores analyzed as they were unable to complete the study due to COVID, this study was terminated.
Time Frame: Enrollment, baseline assessment, 4 weeks of intervention 4-6 times a week, weekly surveys of usability, final assessment; These measures were not completed due to COVID
Population: 0 Caregivers completed their scores on the Vineland Adaptive Behavior Scales, Third Edition, This was due to COVID and not being able to complete the study. This study was terminated. Data were not collected due to early termination of the study.
Groups:
- Caregivers: Caregivers and female and male participants between the ages >3 years and < 9 years of age on date of enrollment from a general population diagnosed with ASD
Arm/Group | Caregivers
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: This study was terminated. no adverse events were not collected due to early termination of the study.
Description: This study was terminated. no adverse events were not collected due to early termination of the study.
Groups:
- Primary: Usability of Cognoa ASD Therapeutic Device
  Zero subjects completed the study due to COVID.
Arm/Group | Primary
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-05-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT04326231/Prot_000.pdf